CLINICAL TRIAL: NCT02273921
Title: EEG Classification System for Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mentis Cura (Industry)
Collaborators: Landspitali University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MC-CT-002
Record Dates: First submitted 2014-09-29; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Dementia
Keywords: Dementia, Diagnosis, Electroencephalography
MeSH Terms: conditions — Dementia; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EEG (No Intervention): A non-invasive EEG recording
  Interventions: Other: EEG recording

INTERVENTIONS:
Other: EEG recording — EEG is recorded once for each participant

SUMMARY:
The goal of this study is to construct a large database of EEG recordings from elderly individuals in predefined groups. The purpose of this database is to select groups of EEG recordings from the database in order to compare the electrophysiology, as measured by EEG, of the groups.

In the clinical trial part all individuals are treated exactly the same and are therefore considered a single group. The categorization is performed during the data analysis.

The groups in the data analysis will initially be based on the following:

1. Healthy controls
2. Mild Cognitive Impairment
3. Alzheimers Disease (AD)
4. Lewy-body Dementia
5. Parkinsons Disease Dementia
6. Vascular Dementia (VaD)
7. Frontotemporal Dementia (FTD)
8. Depression

Other groups will be added if needed.

ELIGIBILITY:
Inclusion Criteria:

* Age of participant in the range of 50-90 years

Exclusion Criteria:

* Outside required age range

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2005-03; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Classification system for dementia based on EEG | The quality of the classification system will be evaluated regularly, at least every 6 months, up to 6 years.
  The EEGs recorded in the trial will be categorized into controls or predefined clinical groups based on the participants' clinical diagnosis. The classification system will be constructed using this categorization.

CONTACTS AND LOCATIONS:
Overall Officials: Jón Snædal, MD, Principal Investigator — Landspitali University Hospital

REFERENCES:
- [Background] Snaedal J, Johannesson GH, Gudmundsson TE, Gudmundsson S, Pajdak TH, Johnsen K. The use of EEG in Alzheimer's disease, with and without scopolamine - a pilot study. Clin Neurophysiol. 2010 Jun;121(6):836-41. doi: 10.1016/j.clinph.2010.01.008. Epub 2010 Feb 12. PMID 20153691
- [Background] Gudmundsson S, Runarsson TP, Sigurdsson S, Eiriksdottir G, Johnsen K. Reliability of quantitative EEG features. Clin Neurophysiol. 2007 Oct;118(10):2162-71. doi: 10.1016/j.clinph.2007.06.018. Epub 2007 Aug 31. PMID 17765604
- [Result] Snaedal J, Johannesson GH, Gudmundsson TE, Blin NP, Emilsdottir AL, Einarsson B, Johnsen K. Diagnostic accuracy of statistical pattern recognition of electroencephalogram registration in evaluation of cognitive impairment and dementia. Dement Geriatr Cogn Disord. 2012;34(1):51-60. doi: 10.1159/000339996. Epub 2012 Aug 23. PMID 22922592